CLINICAL TRIAL: NCT04515524
Title: An Extension Study to Evaluate the Long-Term Outcomes of Patients Who Received Treatment for Retinopathy of Prematurity in the VGFTe-ROP-1920 Study
Brief Title: Extension Study to Evaluate the Long-Term Outcomes of Pediatric Patients Who Received Treatment for Retinopathy of Prematurity in the VGFTe-ROP-1920 Study (Acronym: Butterfleye Next)
Status: Active, not recruiting | Type: Observational
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: VGFTe-ROP-2036; 2020-005875-10 (EudraCT Number); 2024-513231-24-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2020-08-04; First posted 2020-08-17 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ROP patients from VGFTe-ROP-1920: Retinopathy of prematurity (ROP) who were treated with aflibercept and/or laser photocoagulation in study VGFTe-ROP-1920.
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — No study treatment will be administered in this study

SUMMARY:
Primary objectives of the study are:

* To evaluate binocular visual acuity at the end of this study in patients included from the VGFTe-ROP-1920 study, for treatment of Retinopathy of Prematurity (ROP).
* To evaluate long-term safety outcomes in patients included from the VGFTe-ROP-1920 study, for treatment of ROP.

Secondary objectives of the study are:

* To describe visual function in patients included from the VGFTe-ROP-1920 study, for treatment of ROP.
* To describe overall development in patients included from the VGFTe-ROP-1920 study, for treatment of ROP.

ELIGIBILITY:
Inclusion Criteria:

1. Patient was treated in study VGFTe-ROP-1920
2. Age <13 months of chronological age
3. Signed informed consent from parent(s)/legal guardian(s), which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol

Exclusion Criteria:

1. Patient has a condition preventing participation in the study, or performance of study procedures

NOTE: Other Inclusion/Exclusion criteria may apply

Ages: 11 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients who were treated in the VGFTe-ROP-1920 study are eligible for enrollment into this follow-up study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2026-11-05 (Estimated); Study Completion 2026-11-05 (Estimated)

PRIMARY OUTCOMES:
Binocular best-corrected visual acuity (BCVA) | 5 years of chronological age
Proportion of Patients with Adverse Events | Up to 5 years of chronological age
Proportion of Patients with Serious Adverse Events | Up to 5 years of chronological age

SECONDARY OUTCOMES:
Proportion of patients developing unfavorable ocular structural outcome | 3 years of chronological age, 5 years of chronological age
  Unfavorable ocular structural outcome: retinal detachment, macular dragging, macular fold, retrolental opacity
BCVA in each eye | 3 year of chronological age, 5 years of chronological age
Refractive spherical equivalent in each eye | 3 years of chronological age, 5 years of chronological age
Neurodevelopmental outcomes using BSID-III | 2 years of chronological age
  The Bayley Scales of Infant and Toddler Development, Third Edition (BSID-III) is a standard series of tests that will assess the development of children in 3 areas: cognition, language, and motor skills. This is a mandatory assessment to be performed at 2 years of age.
Neurodevelopmental outcomes using WPPSI-IV | 5 years of chronological age
  The Wechsler Preschool and Primary Scale of Intelligence, Fourth Edition (WPPSI-IV) is designed to assess development of older children and is recommended to be performed at 3, 4 and 5 years of age. The assessment at 5 years of age is mandatory. In cases where the WPSSI-IV cannot be used, the Differential Ability Scales II (DAS-II) may be used as an alternative.
Neurodevelopmental outcomes using VABS-II | 2 years of chronological age, 5 years of chronological age
  The Vineland Adaptive Behavior Scales, Second Edition (VABS-II) Expanded Interview will be included, which includes 4 areas: Communication, Daily Living skills, Socialization and Motor Skills. The assessments at 2 years and 5 years of age are mandatory.
Proportion of patients with recurrence of ROP | 3 years of chronological age, 5 years of chronological age
Proportion of patients requiring treatment for ROP | Through 5 years of chronological age

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (30):
- United States (9):
  - UCSD Shiley Eye Institute, Jacobs Retina Center, La Jolla, California
  - Loma Linda University Eye Institute, Loma Linda, California
  - University of California San Francisco - Ophthalmology, San Francisco, California
  - New York University School of Medicine - Oncology, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Lifespan - Women & Infants Hospital of RI, Providence, Rhode Island
  - The Children's Hospital of San Antonio, San Antonio, Texas
  - West Virginia University, Morgantown, West Virginia
- Bulgaria (2):
  - Acibadem City Clinic Multiprofile Hospital for Active Treatment, Sofia
  - Specialized Hospital for Active Treatment of Eye Diseases - Varna, Varna
- Colombia (2):
  - Clinica Universitaria Bolivariana, Medellín, Antioquia
  - Fundacion Oftalmologica de Santander Foscal, Floridablanca, Santander Department
- SC Centrul Medical Unirea SRL, Iași, Romania
- Russia (2):
  - V.F. Voyno-Yasenetsky Scientific and Practical Center of Specialized Medical Care for Children - ophtalmology, Moscow, Moscow
  - St. Petersburg State Pediatric Medical University - ophtalmology, Saint Petersburg
- Soon Chun Hyang University Cheonan Hospital, Cheonan, Chungcheongnam-do, South Korea
- Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan
- Thailand (6):
  - Chulalongkorn University, Bangkok, Bangkok
  - Prince of Songkla University - Ophthalmology, Hat Yai, Changwat Songkhla
  - Phramongkutklao Hospital, Bangkok
  - Queen Sirikit National Institute Of Child Health - Pediatrics, Bangkok
  - Chiang Mai University, Chiang Mai
  - Srinagarind Hospital - Ophthalmology, Khon Kaen
- Turkey (Türkiye) (4):
  - SBU Adana Sehir Training and Research Hospital, Adana
  - Hacettepe University Medical Faculty, Ankara
  - Gazi University Medical Faculty Hospital, Ankara
  - Eskisehir Osmangazi University Medical Faculty Hospital, Eskişehir
- Vietnam (2):
  - Children's Hospital 1 - Ophthalmology Unit, Ho Chi Minh City, Thanh Pho
  - Hue Central Hospital, Huế, Thừa Thiên Huế Province

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/